CLINICAL TRIAL: NCT02060045
Title: Impact of 4 Sequential Measures on the Prevention of Ventilator Associated Pneumonia in Major Heart Surgery Intensive Care Unit
Brief Title: Prevention Ventilator Associated Pneumonia
Acronym: REINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Jesus Perez (Other)
Collaborators: Ciber de Enfermedades Respiratorias (Unknown); Fundación Rafael del Pino (Unknown); Fondo de Investigacion Sanitaria (Other)
Responsible Party: Sponsor-Investigator, Maria Jesus Perez, RN, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: REINA
Record Dates: First submitted 2014-02-04; First posted 2014-02-11 (Estimated); Last update posted 2014-02-11 (Estimated); Status verified 2014-02

CONDITIONS: Ventilator-associated Pneumonia
Keywords: bundle; prevention; Disturbance; Heart, Functional, Postoperative, Cardiac Surgery
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- bundle implementation (Experimental): The measures were a specific training program, aspiration of subglottic secretions (ASS), introduction of an inclinometer to improve the semirecumbent position, and reinforcement of oral care with chlorhexidine.
  Interventions: Other: Bundle implementation

INTERVENTIONS:
Other: Bundle implementation

SUMMARY:
The objective of the investigators work was to evaluate the impact of 4 sequentially implemented measures for preventing VAP in a major heart surgery ICU. The measures were a specific training program, aspiration of subglottic secretions (ASS), introduction of an inclinometer to improve the semirecumbent position, and reinforcement of oral care with chlorhexidine.

ELIGIBILITY:
Inclusion Criteria:

* all patients with heart surgery admitted in critical care unit during the study period

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1534 (Actual)
Dates: Start 2009-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change (reduction) in the incidence density of Ventilator associated pneumonia (VAP) | Baseline and up to 35 months
  Change (reduction) in the incidence density of VAP

SECONDARY OUTCOMES:
Change(length) in Intensive Care Unit (ICU) stay | Baseline and up to 35 months
Change (number of days) in Mechanical Ventilator (MV) per ICU stay | Baseline and up to 35 months
Change in mortality rate | Baseline and up to 35 months
Change in cost of antimicrobial acquisition during ICU stay | Baseline and up to 35 months
Change in compliance with the measures | Baseline and up to 35 months

CONTACTS AND LOCATIONS:
Overall Officials: Maria Jesus Perez, RN, Principal Investigator — Hospital General Universitario Gregorio Marañón
Locations (1):
- Hopsital General Universitario Gregorio Marañon, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Perez-Granda MJ, Barrio JM, Munoz P, Hortal J, Rincon C, Bouza E. Impact of four sequential measures on the prevention of ventilator-associated pneumonia in cardiac surgery patients. Crit Care. 2014 Mar 26;18(2):R53. doi: 10.1186/cc13799. PMID 24667011